CLINICAL TRIAL: NCT00094523
Title: A Phase IIIB/IV, Open-label, Multi-center Trial to Evaluate the Safety, Tolerability, and Efficiency of HIV-1 Infected Subjects Switching Their Current Protease-inhibitor Therapies for a Fosamprenavir Therapy Over 48 Weeks
Brief Title: Fosamprenavir Versus Other Protease Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100290
Record Dates: First submitted 2004-10-20; First posted 2004-10-21 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: fosamprenavir LEXIVA non-inferiority safety tolerability
MeSH Terms: conditions — Infections | interventions — fosamprenavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm A (Experimental): Subjects switched their baseline PI for fosamprenavir (± ritonavir) while maintaining their baseline regimen of two nucleoside or nucleotide reverse transcriptase inhibitors for 48 weeks.
  Interventions: Drug: Fosamprenavir
- Treatment Arm B (Experimental): Subjects continued baseline regimen for first 24 weeks with the option of switching their initial PI for fosamprenavir (± ritonavir) while maintaining their baseline nucleoside or nucleotide reverse transcriptase inhibitor regimen for another 24 weeks
  Interventions: Drug: Fosamprenavir

INTERVENTIONS:
Drug: Fosamprenavir — Fosamprenavir

SUMMARY:
This study was designed to evaluate and compare safety, tolerability of subjects who successfully suppress HIV-1 on their first PI regimen to those who switch to fosamprenavir. This is a 48-week study, where subjects who were assigned to be in their original PI-group have the option of switching to fosamprenavir on week 24. Prior to being assigned their treatment group, subjects had to be suppressed for at least three months. All subjects also take a background regimen of two nucleoside/nucleotide reverse transcriptase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Be on your first protease inhibitor (PI) containing regimen, and the regimen must consist of a PI +/- ritonavir and 2 Nucleoside/Nucleotide Reverse Transcriptase Inhibitors (N[t]RTIs).
* Have a plasma HIV-1 RNA level (viral load) at screening of less than 400 copies/mL, for at least 3 months prior to Screening and at Screening while on your current regimen of a PI +/- ritonavir + 2 N(t)RTIs.
* Females must not be pregnant or breastfeeding or plan to become pregnant during the study.
* Females of child-bearing potential must agree to use one of the approved methods of birth control.

Exclusion Criteria:

* Not able to follow the medication schedules and attend the study visits for the entire length of the study.
* Have any other illnesses, laboratory test results, medication use, allergies, or medical conditions that would make it unsafe for the subject to participate in this study.
* Currently be enrolled in any other research studies that could affect the subject''''s HIV-1 RNA levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2004-12-14 (Actual); Primary Completion 2007-06-29 (Actual); Study Completion 2007-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with HIV-1 RNA less than 400 copies/mL | Week 24

SECONDARY OUTCOMES:
Percentage of subjects with plasma HIV-1 RNA <400 copies/mL | Week 48
Percentage of subjects with plasma HIV-1 RNA <50 copies/mL at Week 24 | Week 24
Percentage of subjects with plasma HIV-1 RNA <50 copies/mL at Week 48 | Week 48
Number of subjects with any adverse events (AEs) | up to Week 48
Number of subjects with gastrointestinal (GI) AEs | up to Week 48
Absolute values of plasma HIV-1 RNA at Week 24 | Week 24
Median change from Baseline in HIV-1 RNA at Week 24 | Baseline and Week 24
Absolute values of plasma HIV-1 RNA at Week 48 | Week 48
Median change from Baseline in HIV-1 RNA at Week 48 | Baseline and Week 48
Absolute values in Cluster of Differentiation 4+ (CD4+) Cell Counts at Week 24 | Week 24
Absolute values in Cluster of Differentiation 4+ (CD4+) Cell Counts at Week 48 | Week 48
Median change from Baseline in Cluster of Differentiation 4+ (CD4+) Cell Counts at Week 24 | Baseline and Week 24
Median change from Baseline in Cluster of Differentiation 4+ (CD4+) Cell Counts at Week 48 | Baseline and Week 48
Number of subjects with genotypic resistance at virologic failure | up to Week 48
Number of subjects with phenotypic resistance at virologic failure | up to Week 48
Time to loss of virologic response (TLOVR) | up to Week 48
Medication adherence at Week 24 | Week 24
Medication adherence at Week 48 | Week 48
Subject treatment satisfaction per the HIV Treatment Satisfaction Questionnaire at Week 24 | Week 24
Subject treatment satisfaction per the HIV Treatment Satisfaction Questionnaire at Week 48 | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (46):
- United States (45):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Laguna Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Morristown, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Hampton, Virginia
- GSK Investigational Site, Ponce, Puerto Rico